CLINICAL TRIAL: NCT05641259
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of LP-108, a BCL-2 Inhibitor, Combined With Azacitidine In Subjects With AML, MDS, CMML
Brief Title: A Study to Assess Safety and Preliminary Efficacy of LP-108 Combined With Azacitidine In Subjects With AML, MDS, CMML
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Guangzhou Lupeng Pharmaceutical Company LTD. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LP-108-CN102
Record Dates: First submitted 2022-11-17; First posted 2022-12-07 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes; Chronic Myelomonocytic Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic | interventions — Azacitidine

STUDY DESIGN:
Intervention Model Description: This is a Phase 1 study with a dose escalation design and an expansion cohort.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dose Escalation (Experimental): LP-108: Cycle 0: ramp-up from Day 1, Cycle 1+: at escalating dose levels in participants with AML, MDS or CMML.
  Azacitidine: beginning on Day 1 through Day 7 of each Cycle (expect for Cycle 0).
  Strong/moderate CYP3A inhibitor and inducer are prohibited. Participants are treated indefinitely until disease progression, unacceptable toxicity or withdrawal for other reasons.
  Interventions: Drug: LP-108; Drug: Azacitidine
- Safety Expansion (Experimental): LP-108: Cycle 0: ramp-up from Day 1, Cycle 1+: Participants with AML, MDS or CMML will be treated with LP-108 to enable selection of the recommended Phase 2 dose (RP2D).
  Azacitidine: beginning on Day 1 through Day 7 of each Cycle (expect for Cycle 0).
  Strong/moderate CYP3A inhibitor and inducer are prohibited. Participants are treated indefinitely until disease progression, unacceptable toxicity or withdrawal for other reasons.
  Interventions: Drug: LP-108; Drug: Azacitidine
- Efficacy Expansion [AML] (Experimental): LP-108: Cycle 0: ramp-up from Day 1, Cycle 1+: at RP2D level in participants with AML .
  Azacitidine: beginning on Day 1 through Day 7 of each Cycle (expect for Cycle 0).
  After the completion of Part 1, the Part 2 dose expansion phase will begin. Strong/moderate CYP3A inhibitor and inducer are prohibited. Participants are treated indefinitely until disease progression, unacceptable toxicity or withdrawal for other reasons.
  Interventions: Drug: LP-108; Drug: Azacitidine
- Efficacy Expansion [MDS&CMML] (Experimental): LP-108: Cycle 0: ramp-up, Cycle 1+: at RP2D level in participants with MDS or CMML.
  Azacitidine: beginning on Day 1 through Day 7 of each Cycle (expect for Cycle 0).
  Strong/moderate CYP3A inhibitor and inducer are prohibited. Participants are treated indefinitely until disease progression, unacceptable toxicity or withdrawal for other reasons.
  Interventions: Drug: LP-108; Drug: Azacitidine

INTERVENTIONS:
Drug: LP-108 — Oral administration for 21 or 28 days on a 28-day cycle
Drug: Azacitidine — Subcutaneous administration for 7 days on a 28-day cycle at the dose of 75mg/m2 2-2.5h hours after LP-108.

SUMMARY:
This is a Phase 1, open-label, multicenter, dose-escalation & expansion study to evaluate the safety,tolerability and pharmacokinetics (PK) of LP-108, a BCL-2 inhibitor, combined with azacitidine, to determine the dose limiting toxicity (DLT) and the recommended Phase 2 dose (RP2D), and to assess the preliminary efficacy of this combination.

DETAILED DESCRIPTION:
This Phase 1 study will look at different doses and different treatment schedules in order to better understand the effects of the combined regimens on the newly diagnosed or refractory/relapsed adult participants with AML ,MDS or CMML. The procedures include screening for eligibility, study treatments, and blood & bone marrow tests. All the safety events will be record, pharmacokinetic parameters (Tmax, Cmax,T1/2, AUC et al.) will be calculated, response and survival will be assess during the study. Participants will be treated indefinitely until disease progression, unacceptable toxicity or withdrawal for other reasons.

ELIGIBILITY:
Inclusion Criteria:

* Subject must has a diagnosis of one of the following: relapsed or refractory (R/R) or untreated ineligible for treatment with a standard induction chemotherapy acute myeloid leukemia (AML) ; R/R myelodysplastic syndrome(MDS) or untreated MDS with excess blasts defined as ≥ 5% blasts in either bone marrow or blood or with high risk (high and very high-risk groups according to IPSS-R) ;CMML-1 or 2 by WHO, no requirements for prior therapy.
* ECOG performance status ≤ 2.
* Estimated survival ≥ 12 weeks.
* Baseline white blood cell count (WBC) ≤ 25 x 109/L.
* Subject must has adequate organ function as defined below: Aspartate transaminase (AST) and alanine transaminase (ALT)≤3 x ULN; Bilirubin ≤1.5 x ULN (unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin); adequate renal function as demonstrated by a creatinine clearance ≤1.5 x ULN ; calculated by the Cockcroft Gault formula; APTT ≤ 1.5 x ULN, INR ≤ 1.5 x ULN.
* Prior treatment-related toxicities must be grade 1 or baseline except for alopecia.
* If subject is sexually active, he/she must agree to carry out birth control throughout the study and 90 days after the last dose of LP-108. Subject must agree to have a negative serum β-HCG test result within 7 days prior to study drug.
* Subject must voluntarily sign and date an informed consent.

Exclusion Criteria:

* Subject is allergic to LP-108, Azacitidine or excipients, or with poor tolerance to Azacitidine.
* Subject has received prior therapy with a BH3 mimetic.
* Subject has acute promyelocytic leukemia.
* Subject has t(9;22) karyotype abnormality or positive BCR/ABL1 fusion gene.
* Subject has known and active CNS involvement.
* Subject has myeloid sarcoma but no bone marrow involvement.
* Subject has Acute unidentified leukemia.
* Subject has treatment related MDS or AML.
* Subject has AML/MDS/CMML with myelofibrosis ≥ grade 2.
* Subject has received allogeneic Hematopoietic Stem Cell Transplantation (HSCT) or autologous HSCT within 3 months prior to the first dose of study drug.
* Subject must be at least 4 weeks from antitumor therapy, major surgery, radiation therapy, or participation in other investigational trials.
* Subject has received a strong and/or moderate CYP3A inhibitor or inducer, P-gp inhibitor or CYP2C8 substrate within 14 days prior to the initiation of study treatment.
* Subject has received drugs with a potential to cause prolonged QT intervals or torsade de pointes.
* Administration or consumption of any of the following within 3 days prior to the first dose of study drug: Grapefruit or grapefruit products; Seville oranges (including marmalade containing Seville oranges); Star fruit.
* Subject has known malignancy within 3 years prior to the first dose of study drug, with the exception of: Adequately treated basal skin cancers, in situ carcinoma of the cervix uteri or breast, localized squamous cell carcinoma.
* Subject has serious and/or uncontrolled systemic diseases, in the opinion of the investigator, the subject is inappropriate for enrollment into this study (serious active infection with grade ≥ 2(based on CTCAE), high blood pressure that cannot be controlled by medication, diabetes, unstable angina, congestive heart failure, Respiratory diseases requiring continuous oxygen intake, severe vascular embolism, uncontrolled massive bleeding or bleeding from vital organs, severe liver, kidney or metabolic diseases, such as cirrhosis, kidney failure, etc.).
* Subject has myocardial infarction or stroke within 6 months prior to the first dose of study drug.
* Subject has a cardiac history including the following: History of CHF requiring treatment or Ejection Fraction <50% or a cardiovascular disability status of New York Heart Association.
* Subject has uncontrolled and/or active systemic infection (viral, bacterial or fungal).
* Subject has difficulty to swallow pills or has conditions that affect drug absorption or pharmacokinetics.
* Strong and/or moderate CYP3A inhibitor or inducer and CYP2C8 substrate cannot be discontinued during the study.
* Vaccination with live, attenuated vaccines ≤4 weeks prior to initiation of study treatment or anticipation of need for such a vaccine during the study or 4 weeks after the last dose of study drug.
* Subject has an autoimmune disease that requires immunosuppressive therapy In the opinion of the investigator, the subject is inappropriate for enrollment into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2023-02-14 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose(MTD) | Up to 42 days after initial dose of study drug at the designated cohort dose.
  Standard phase I 3+3 design. The first 3 subjects will be assigned to dose level 1 cohort. If none of the first three subjects experiences DLT, escalation to dose level 2 cohort is permitted. If one of the first three subjects' experiences DLT, a total of six subjects will be required in that dose cohort, and escalation will only be permitted if five of six subjects do not experience DLT. If more than one DLT is observed in the dose level 2 cohort, this will be determined to be the maximally administered dose, and three more subjects will be enrolled in the dose level 1 cohort if only three were previously treated at that dose. Escalation from dose level 2 to level 3 cohort will be with the same method as before. The MTD will be the cohort in which ≤1/6 subjects have dose limiting toxicity at the dose prior to the maximally administered dose. If the dose level 3 cohort has ≤1/6 subjects with a DLT, the MTD will not have been reached.
Recommended Phase 2 Dose(RP2D) | Up to 1.5 years
  RP2D will be determined using available safety and pharmacokinetics data upon completion of the dose escalation phase.
Incidence of AEs | From first dose of study drug to 28 days after last dose of study drug
  Type, frequency and severity of AEs, relationship of AEs to study treatment
Incidence of clinically significant changes in clinical laboratory results | From first dose of study drug to 28 days after last dose of study drug
  Clinically significant changes in hematology, chemistry, coagulation and urinalysis tests results.
Cmax of LP-108 | Up to 24 hours post dose
  Maximum plasma concentration (Cmax) of LP-108.
Tmax of LP-108 | Up to 24 hours post dose
  Time to maximum plasma concentration (Tmax) of LP-108.
t1/2 of LP-108 | Up to 24 hours post dose
  The terminal elimination half-life (t1/2).
AUC0-t of LP-108 | Up to 24 hours post dose
  Area under the plasma concentration-time curve (AUC) from 0 to the time of the last measurable concentration of LP-108.
CL/F of LP-108 | Up to 24 hours post dose
  Apparent clearance (CL/F) of LP-108.
Vd/F of LP-108 | Up to 24 hours post dose
  Apparent volume of distribution of LP-108.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Measured from Cycle 1 Day 1 to 28 days after last dose of study drug, and assessed up to 24 months.
  Response criteria follows the 2017 European Leukemia Net (ELN) recommendations for AML( CR, CRi, PR) , the International Working Group (IWG) response criteria for MDS(CR, PR, marrow CR, HI), the international consortium proposal of uniform response criteria for myelodysplastic/myeloproliferative neoplasms (MDS/MPN) in adults(CR, PR, Marrow response, Clinical benefit).
Progression-Free Survival(PFS) (only for MDS or CMML) | Measured from the date of first dose of study drug to the date of earliest disease progression or death or last visit, and assessed up to 24 months.
  PFS is defined as the number of days from the date of the first dose of study drug to the date of earliest disease progression or death.
Time to Response(TTR) | Measured from the date of the first dose of study drug to the date of earliest response, and assessed up to 6 months.
  TTR is defined as the number of days from the date of the first dose of study drug to the date of earliest response.
Duration of Response(DOR) | Measured from the date of the first remission to the date of earliest disease progression or death, and assessed up to 24 months.
  DOR is defined as the number of days from the date of the first remission to the date of earliest disease progression or death.
DOCR (only for CR/CRi participants) | Measured from the date of the first CR/CRi to the date of earliest disease progression or death, and assessed up to 24 months.
  DOCR is defined as the number of days from the date of the first CR/CRi to the date of earliest disease progression or death.
Event-free Survival (EFS) | Measured from the date of first dose to the date of earliest evidence of disease progression, initiation of new non-protocol-specified antitumor therapy without documented progression, death, and for up to 5 years after the last subject is enrolled.
  EFS is defined as the number of days from the date of first dose to the date of earliest evidence of disease progression/relapse, or initiation of new non-protocol-specified antitumor therapy without documented progression, or death.
OS | Measured from the date of date of first dose to the date of death or last visit, and for up to 5 years after the last subject is enrolled.
  OS is defined as the number of days from the date of first dose to the date of death.

CONTACTS AND LOCATIONS:
Overall Officials: Depei Wu, PhD, Study Chair — First Affiliated Hospital of Soochow University; Xudong Wei, PhD, Principal Investigator — Affiliated Tumor Hospital of Zhengzhou University, Henan Cancer Hospital; Qiubai Li, PhD, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology; Li Wang, PhD, Principal Investigator — First Affiliated Hospital of Chongqing Medical University; Fei Li, PhD, Principal Investigator — The First Affiliated Hospital of Nanchang University; Xiaojing Yan, PhD, Principal Investigator — First Hospital of China Medical University
Locations (3):
- China (3):
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - First Affiliated Hospital of Soochow University, Suzhou
  - Affiliated Tumor Hospital of Zhengzhou University, Henan Cancer Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dohner H, Estey E, Grimwade D, Amadori S, Appelbaum FR, Buchner T, Dombret H, Ebert BL, Fenaux P, Larson RA, Levine RL, Lo-Coco F, Naoe T, Niederwieser D, Ossenkoppele GJ, Sanz M, Sierra J, Tallman MS, Tien HF, Wei AH, Lowenberg B, Bloomfield CD. Diagnosis and management of AML in adults: 2017 ELN recommendations from an international expert panel. Blood. 2017 Jan 26;129(4):424-447. doi: 10.1182/blood-2016-08-733196. Epub 2016 Nov 28. PMID 27895058
- [Result] Cheson BD, Greenberg PL, Bennett JM, Lowenberg B, Wijermans PW, Nimer SD, Pinto A, Beran M, de Witte TM, Stone RM, Mittelman M, Sanz GF, Gore SD, Schiffer CA, Kantarjian H. Clinical application and proposal for modification of the International Working Group (IWG) response criteria in myelodysplasia. Blood. 2006 Jul 15;108(2):419-25. doi: 10.1182/blood-2005-10-4149. Epub 2006 Apr 11. PMID 16609072
- [Result] Savona MR, Malcovati L, Komrokji R, Tiu RV, Mughal TI, Orazi A, Kiladjian JJ, Padron E, Solary E, Tibes R, Itzykson R, Cazzola M, Mesa R, Maciejewski J, Fenaux P, Garcia-Manero G, Gerds A, Sanz G, Niemeyer CM, Cervantes F, Germing U, Cross NC, List AF; MDS/MPN International Working Group. An international consortium proposal of uniform response criteria for myelodysplastic/myeloproliferative neoplasms (MDS/MPN) in adults. Blood. 2015 Mar 19;125(12):1857-65. doi: 10.1182/blood-2014-10-607341. Epub 2015 Jan 26. PMID 25624319